CLINICAL TRIAL: NCT01259245
Title: Effectiveness of Incorporating Tai Chi in Pulmonary Rehabilitation Program for COPD Patients in Primary Health Care
Brief Title: Effectiveness of Incorporating Tai Chi in Pulmonary Rehabilitation Program for Chronic Obstructive Pulmonary Disease Patients in Primary Health Care
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Lorna Ventura Ng, Senior Medical Officer, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHSRF08091291
Record Dates: First submitted 2010-12-03; First posted 2010-12-14 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease COPD; pulmonary rehabilitation program PRP; Tai chi
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai chi + PRP (Experimental): Tai chi elements in incorporated into the exercise component of standard pulmonary rehabilitation program. The exercise content was totally identical to the PRP group except 15 minutes of Tai Chi exercises was substituted to 15 minutes of relaxation exercise. The 5 forms of Sun Style of Tai Chi were taught.
  Interventions: Other: Tai chi + PRP; Other: PRP
- PRP (Active Comparator): PRP is a formal pulmonary rehabilitation program consisted of physical training including warm up and cool down exercise and aerobic exercises in addition to breathing control exercises, safety precautions for physical training, Thera-Band strengthening exercises and overview of COPD management.
  Interventions: Other: PRP

INTERVENTIONS:
Other: Tai chi + PRP — The exercise content was totally identical to PRP group except 15 minutes of 5 Sun Style Tai Chi were substituted to 15 minutes of relaxation exercise
  Other Names: Tai chi elements added to pulmonary rehabilitation program
  Arms: Tai chi + PRP
Other: PRP — Formal pulmonary rehabilitation program consisted of overview of COPD management, aerobic exercises, breathing control exercises, Thera-Band strengthening exercises, safety precautions for physical training and goal setting
  Other Names: Formal pulmonary rehabilitation program

SUMMARY:
The purpose of this study was to compare the self-efficacy and quality of life parameters of Chronic Obstructive Pulmonary Disease(COPD)patients who underwent pulmonary rehabilitation with and without Tai Chi elements incorporated in the exercise component in a General Out-patient setting.

DETAILED DESCRIPTION:
Subjects: 192 patients were enrolled and recruited from four General Out-patient clinics in Yau Tsim Mong and Wong Tai Sin districts.

Study Design: Prospective single blind randomized controlled trial

Subjects were randomized into Pulmonary rehabilitation program (PRP) group (n = 98) and Pulmonary rehabilitation program with Tai chi group (TC)(n=94). Details of PRP and PRP + Tai Chi will be discussed below.

Both groups will be given booklet on COPD information and management.

Randomization:

Computer generated pre-assigned randomization of subjects to group allocation is made after baseline assessment. At each stage, assessors for outcome measures and data collection are blinded to the patient's grouping. Patients, investigator and physiotherapist are open to the group allocation.

Standardized medical treatment:

All COPD patients are managed according to practical guidelines recommended by the Hospital Authority. Medical treatment is reviewed and changed if clinically appropriate. In response to an exacerbation, antibiotic is added if a respiratory infection is the cause and oral steroid may be prescribed if clinically indicated.

Measurement and Evaluation

Baseline assessment:

1. Medical aspect: GOLD staging of COPD; Baseline spirometry test including bronchodilator reversibility test.
2. Self-Efficacy: COPD Self Efficacy Scale (CSES); Self-Efficacy for Managing Shortness of Breath (SEMSOB)
3. Quality of life related measures: St. George Respiratory Questionnaire ( SGRQ)
4. Exercise Capacity: 6 Minutes Walking Distance Test (6MWT)

Reassessment done at 2 months and 6 months using:

1. Primary Outcome measures and Secondary measures outcome mentioned in outcome measures
2. Spirometry exclusive of bronchodilator reversibility test

Statistical methods

Descriptive statistics including mean, standard deviation, frequency and percentages were used to describe the demographic characteristics and summarize the baseline characteristics of the variables. Independent T-test was used to examine the difference in demographic characteristics and baseline outcome measures between the PRP and TC group. Paired T-test was performed to examine the differences of outcome measures, including spirometry, 6 MWT, SGRQ-HKC, CSES, SEMSOB before and after intervention program within group. Analysis of covariance(ANCOVA) were used to examine the differences of outcome variables between PRP and TC group adjusted for age, sex, body mass index BMI, smoking and education, with the corresponding baseline value as a covariate. A p-value of 0.05 ws used as the level of statistical significance. Confidence intervals ( 95%) of the mean differences between baseline and 6 months post intervention values were calculated to compare the effects with the minimum clinically important difference (MCID) for the SGRQ-HKC. All analyses were conducted using Statistical package for the Social Sciences SPSS version 16.0.

Pulmonary Rehabilitation Programme (PRP) Details :

The revised PRP consisted of 12 sessions (twice per week for 6 weeks) with 6-10 subjects per session. The standard content consists of physical training including warm up & cool down exercise and aerobic exercises.

For the PRP group, patients performed 5 minutes warm up exercises. Then 2 aerobic activities including treadmill exercise and lower limb ergometry exercise lasting 20 minutes each,were prescribed. 15 minutes rest were given between each exercise. After the aerobic exercises, 5 minutes cool down exercises, followed by 15 minutes of relaxation exercise was conducted before patients completed that session. Each session lasted for about 1 hour and 20 minutes.They were instructed to continue unsupervised home exercises consisting of 5 minutes of warm-up, 5 minutes of Thera-Band strengthening exercises, 30 minutes of aerobic exercises, 5 minutes cool down and 15 minutes of relaxation exercise for at least one hour 5-7 days/week.

For the PRP + Tai Chi group, the exercise content is totally identical to the PRP group except 15 minutes of Tai Chi exercises was substituted to the 15 minutes of relaxation exercise. Each session also lasted for about 1 hour and 20 minutes. The 5 forms of Suen Style of Tai Chi are chosen because it will encourage larger limbs movement as well as chest wall movement incorporated with diaphragmatic breathing and breathing control.

Details of the 5 forms of Sun Style Tai Chi chosen are:

1. commencing form
2. single whip : left and right
3. turn with slanted flying: left and right
4. wave hands like clouds: left and right
5. moving as if shutting a door

The exercise intensity level of the aerobic activities will be set at a target heart rate of 60-70 % of their maximum heart rate and rate of perceived dyspnea(RPD) level of not more than 7. Vital signs will be monitored before, during & after exercise to ensure that the exercise heart rate does not exceed the target level. Also, any time when patient feels discomfort with RPD level reaching 7, the exercise will be stopped and patient is allowed to rest.

ELIGIBILITY:
Inclusion Criteria:

1. . Previous diagnosis of COPD
2. . Absence of bronchiectasis, bronchiolitis obliterans, panbronchiolitis and asthma
3. . Medical Research Council(MRC)Dyspnea score > 2 using the 1-5 scale version
4. .Willing to participate and able to give consent

Exclusion Criteria:

1. . Patients with poor mobility, i.e. wheelchair bound; or
2. . Patients with severe comorbidities, including acute myocardial infarction in preceding 6 months; or
3. . Patients with severe hearing impairment or cognitive impairment; or
4. . Patient unwilling to participate and unable to give consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: lorna Ng, doctor, Principal Investigator — Kwong Wah Hospital
Locations (1):
- Kwong Wah Hospital General Out-patient Clinic, Hong Kong SAR, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment and intervention part of the study took place between March 2011 and November 2011 with follow-up until May 2012. Subjects were recruited from four difference general out-patient clinics (GOPCs.
Pre-assignment Details: Using the inclusion and exclusion criteria, 192 adult subjects were enrolled into the study
Groups:
- Pulmonary Rehabilitation Program: PRP is a formal pulmonary rehabilitation program consisted of physical training including warm up and cool down exercise and aerobic exercises in addition to breathing control exercises, safety precautions for physical training, Thera-Band strengthening exercises and overview of COPD management.
  PRP : Formal pulmonary rehabilitation program consisted of overview of COPD management, aerobic exercises, breathing control exercises, Thera-Band strengthening exercises, safety precautions for physical training and goal setting
- Tai Chi + PRP: Tai chi elements in incorporated into the exercise component of standard pulmonary rehabilitation program. The exercise content was totally identical to the PRP group except 15 minutes of Tai Chi exercises was substituted to 15 minutes of relaxation exercise. The 5 forms of Sun Style of Tai Chi were taught.
  PRP : Formal pulmonary rehabilitation program consisted of overview of COPD management, aerobic exercises, breathing control exercises, Thera-Band strengthening exercises, safety precautions for physical training and goal setting
  Tai chi + PRP : The exercise content was totally identical to PRP group except 15 minutes of 5 Sun Style Tai Chi were substituted to 15 minutes of relaxation exercise
Period: Overall Study
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Started | 98 | 94
Completed | 70 (27 were lost to follow-up and 1 deceased) | 68 (24 discontinued intervention and 2 deceased)
Not Completed | 28 | 26
Not completed — Withdrawal by Subject | 27 | 24
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP | Total
Number analyzed (Participants) | 98 | 94 | 192
Age Continuous [Mean (Standard Deviation); unit: years] | 74 (6.81) | 74 (6.41) | 74 (6.624)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 87 | 88 | 175
Region of Enrollment [Number; unit: participants]
  Hong Kong | 98 | 94 | 192
COPD-CSES [Mean (Standard Deviation); unit: rating score 0.2 to 1] — COPD Self-efficacy scale is a 34-item questionnaire which measures a person's confidence in managing or avoiding breathing difficulties in a number of situations categorized under 5 factors or condition. It consists of Likert scale with 5 responses ranging from "1" -not at all confident" to "5" - very confident" with higher scores representing higher self efficacy. In this study, a rating score which takes account of items that may not be applicable to the patient by reporting the average score based on the number of items answered. Minimum score 0.2 to maximum score of 1(higher self-efficacy)
  rating score 0.2 to 1 | 0.684 (0.165) | 0.638 (0.152) | 0.661 (0.160)
SEMSOB [Mean (Standard Deviation); unit: likert scale] — Self-efficacy for managing shortness of breath is a single question 1-10 scale, valid and reliable instrument that measures patients' overall confidence in keeping breathing difficulties from interfering with what they want to do with higher score indication greater self efficacy.
  likert scale | 6.86 (2.34) | 6.53 (1.98) | 6.70 (2.171)
SGRQ HKC Symptom [Mean (Standard Deviation); unit: score from 0 to 100] — The Saint George Respiratory Questionnaire (SGRQ HKC) is a Hong Kong Chinese validated version of a disease specific measure of health status applicable for use in COPD patients. It consists of 50 items with 76 weighted responses and has three component scores: symptoms, activity and impact. SGRQ HKC Symptom score is calculated by dividing the summed weights by adjusted maximum possible weight for that component and expressing the result as a percentage. SGRQ-Symptom score ranged from 0 to 100, where zero indicates best health and 100 indicating maximum disability.
  score from 0 to 100 | 27.57 (19.71) | 29.77 (19.94) | 28.65 (19.80)
SGRQ HK-Activity [Mean (Standard Deviation); unit: score from 0 to 100] — The Saint George Respiratory Questionnaire (SGRQ HKC) is a Hong Kong Chinese validated version of a disease specific measure of health status applicable for use in COPD patients.It consists of 50 items with 76 weighted responses and has three component scores: symptoms, activity and impact. SGRQ HKC-Activity score is calculated by dividing the summed weights by adjusted maximum possible weight for that component and expressing the result as a percentage. Score ranged from 0 to 100, where zero indicates best health and 100 indicating maximum disability.
  score from 0 to 100 | 43.08 (23.42) | 50.75 (22.77) | 46.84 (23.36)
SGRQ HKC-Impact [Mean (Standard Deviation); unit: score from 0 to 100] — The Saint George Respiratory Questionnaire (SGRQHKC) is a Hong Kong Chinese validated version of a disease specific measure of health status applicable for use in COPD patients. It consists of 50 items with 76 weighted responses and has three component scores: symptoms, activity and impact. SGRQ HKC-Impact score is calculated by dividing the summed weights by adjusted maximum possible weight for that component and expressing the result as a percentage. Score ranged from 0 to 100, where zero indicates best health and 100 indicating maximum disability.
  score from 0 to 100 | 24.11 (17.37) | 27.43 (20.02) | 25.74 (18.74)
SGRQ-HKC Total [Mean (Standard Deviation); unit: score from 0 to 100] — SGRQ HKC-total is the total score calculated from all three components (Symptom, activity and impact)by summing all positive responses in the questionnaire and expressing the result as a percentage of the total weight for the questionnaire. SGRQ total score also range from 0 to 100, where zero indicates best health and 100 indicating maximum disability.
  score from 0 to 100 | 30.44 (17.16) | 34.89 (18.39) | 32.61 (17.87)
6 MWT [Mean (Standard Deviation); unit: Distance in meters] — The 6 minute walking distance test measured the self paced distance that a patient could quickly walk on a flat, hard surface in a period of 6 minutes.
  Distance in meters | 320.2 (71.86) | 312.1 (64.15) | 316.22 (68.14)
FVC [Mean (Standard Deviation); unit: liters] — Forced vital capacity is a component of lung function parameters measured using spirometry
  liters | 2.26 (0.80) | 2.05 (0.66) | 2.15 (0.74)
FEV1 [Mean (Standard Deviation); unit: liters] — Forced expiratory volume in one second ; component of lung function parameters measured by spirometry
  liters | 1.23 (0.45) | 1.10 (0.45) | 1.16 (0.46)
FEV1% Pred [Mean (Standard Deviation); unit: percentage of predicted normal values] — Pred FEV1 percent predicted normal values ; component of lung function parameters measured by spirometry
  percentage of predicted normal values | 63.1 (22.11) | 56.38 (23.81) | 59.82 (23.15)

OUTCOME MEASURES:

1. Primary Outcome: Self Efficacy :COPD Self Efficacy Scale (CSES)
Description: 34 item questionnaire consisting of likert scale with 5 responses ranging from "1" indicating " not at all confident" to "5" indicating " very confident" with higher scores representing higher self efficacy. In this study , we used the rating score in the analysis as some items were considered non-applicable in some cases. Rating score from 0.2 to 1 with 0.2 as "not at all confident and 1 as "very confident". The validated Chinese version of CSES was also used
Time Frame: Change in CSES at 6 months post-intervention
Population: Intention to treat was used in the analysis
Measure: Mean (Standard Deviation); unit: rating score of 0.2 to 1
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Number analyzed (Participants) | 98 | 94
rating score of 0.2 to 1 | 0.733 (0.143) | 0.685 (0.137)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs Tai Chi + PRP; Test type: Superiority or Other; p = 0.252, ANCOVA — Regression coefficients from ANCOVA for Tai Chi intervention (PRP as reference) at 6 months after adjusted for baseline value of the outcome variable, age, sex, BMI, smoking and education; Mean Difference (Final Values) = -0.017, 95% CI 2-sided [-0.046 to 0.012]

2. Primary Outcome: Self- Efficacy : Self-Efficacy for Managing Shortness of Breath ( SEMSOB)
Description: The SEMSOB is a single question 1-10 scale, valid and reliable instrument that measures patients' overall confidence in keeping breathing difficulties from interfering with what they want to do with higher score indicating greater self efficacy.
Time Frame: Change in SEMSOB at 6 months post-intervention
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation Program | PRP+Tai Chi
Number analyzed (Participants) | 98 | 94
units on a scale | 7.13 (1.98) | 7.03 (1.75)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs PRP+Tai Chi; power0.80 for a medium effect size at 5% level of significance; Test type: Superiority or Other; p = 0.984, ANCOVA; Adjusted for baseline values, age, sex, education, BMI and smoking; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.438 to 0.447], Standard Deviation 0.442

3. Primary Outcome: SGRQ HKC-Symptoms
Description: SGRQ HKC-Symptoms is calculated by dividing the summed weights by the adjusted maximum possible weight for that component and expressing the result as a percentage. SGRQ-Symptoms score ranged from 0 to 100, where zero indicates best health and 100 indicating maximum disability.
Time Frame: 6 months post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Number analyzed (Participants) | 98 | 94
units on a scale | 23.49 (19.53) | 25.58 (20.06)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs Tai Chi + PRP; power of 0.80 for a medium effect size at 5% level of significance; Test type: Superiority or Other; p = 0.869, ANCOVA; adjusted for baseline values, age, sex, education, BMI and education; Mean Difference (Final Values) = 0.372, 95% CI 2-sided [-4.061 to 4.805], Standard Deviation 4.433

4. Primary Outcome: SGRQ HKC-Activity
Description: SGRQ HKC-Activity is calculated by dividing the summed weights by the adjusted maximum possible weight for that component and expressing the result as a percentage. SGRQ-Activity score from 0 to 100, where zero indicates best health and 100 indicating maximum disability.
Time Frame: 6 months post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Number analyzed (Participants) | 98 | 94
units on a scale | 41.04 (21.84) | 44.92 (21.89)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs Tai Chi + PRP; power of 0.80 for medium size effect at 5% level of significance; Test type: Superiority or Other; p = 0.588, ANCOVA; adjusted for baseline values, age, sex, BMI, education and smoking; Mean Difference (Final Values) = -1.295, 95% CI 2-sided [-6.001 to 3.411], Standard Deviation 4.706

5. Primary Outcome: SGRQ HKC-Impact
Description: SGRQ HKC -Impact is calculated by dividing the summed weights by the adjusted maximum possible weight for that component and expressing the result as a percentage. SGRQ-impact score from 0 to 100, where zero indicates best health and 100 indicating maximum disability.
Time Frame: 6 months post-intervention
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Number analyzed (Participants) | 98 | 94
units on a scale | 19.56 (19.36) | 20.23 (19.27)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs Tai Chi + PRP; power of 0.80 for medium effect size at 5% level of significance; Test type: Superiority or Other; p = 0.345, ANCOVA; adjusted for baseline values, age, sex, BMI, education and smoking; Mean Difference (Final Values) = -2.150, 95% CI 2-sided [-6.627 to 2.327], Standard Deviation 4.477

6. Primary Outcome: SGRQ HKC Total
Description: SGRQ HKC-Total is calculated by summing all positive responses in the questionnaire and expressing the result as a percentage of the toal weight for the questionnaire. A total score is calculated from all three components. The SGRQ-total score ranged from 0 to 100, where zero indicates best health and 100 indicating maximum disability.
Time Frame: 6 months post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Number analyzed (Participants) | 98 | 94
units on a scale | 26.72 (18.39) | 28.60 (18.33)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs Tai Chi + PRP; power of 0.80 for medium effect size at 5% level of significance; Test type: Superiority or Other; p = 0.413, ANCOVA; adjusted for baseline value, age, sex, BMI, education and smoking; Mean Difference (Final Values) = -1.690, 95% CI 2-sided [-5.753 to 2.372], Standard Deviation 4.062

7. Secondary Outcome: 6 MWT in Meters
Description: The 6 minute walking test ( 6MWT) was conducted according to protocol recommended by American Thoracic Society (ATS) guidelines to measure functional exercise capacity.This test measured the self paced distance in meters that a patient could quickly walk on a flat, hard surface in a period of 6 minutes.
Time Frame: 6 months post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Number analyzed (Participants) | 98 | 94
meters | 335.1 (68.49) | 340.2 (74.20)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs Tai Chi + PRP; power of 0.80 for medium effect size at 5% level of significance; Test type: Superiority or Other; p = 0.004, ANCOVA; adjusted for baseline value, age, sex, BMI, education and smoking; Mean Difference (Final Values) = 13.049, 95% CI 2-sided [4.159 to 21.939], Standard Deviation 8.89

8. Secondary Outcome: FVC
Description: Forced vital capacity, measured in liters, component of lung function parameters measured by spirometry
Time Frame: 6 months post intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Number analyzed (Participants) | 98 | 94
liters | 2.26 (0.77) | 2.18 (0.75)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs Tai Chi + PRP; power of 0.80 for medium effect size at 5% level of significance; Test type: Superiority or Other; p = 0.560, ANCOVA; adjusted for baseline value, age, sex, BMI, education and smoking; Mean Difference (Final Values) = 0.042, 95% CI 2-sided [-0.100 to 0.184], Standard Deviation 0.226

9. Secondary Outcome: FEV1
Description: Forced expiratory volume in one second, measured in liters, component of lung function test measured by spirometry
Time Frame: 6 months post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Number analyzed (Participants) | 98 | 94
liters | 1.28 (0.51) | 1.21 (0.52)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs Tai Chi + PRP; power of 0.80 for medium effect size at 5% level of significance; Test type: Superiority or Other; p = 0.425, ANCOVA; adjusted for baseline value, age, sex, BMI, education and smoking; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [-0.054 to 0.128], Standard Deviation 0.088

10. Secondary Outcome: FEV1% Pred
Description: Pred FEV1 percent predicted normal values;measured using spirometry
Time Frame: 6 months post-intervention
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of FEV1 predicted
Arm/Group | Pulmonary Rehabilitation Program | Tai Chi + PRP
Number analyzed (Participants) | 98 | 94
percentage of FEV1 predicted | 66.2 (24.75) | 62.52 (27.65)
Statistical Analysis 1: Comparison: Pulmonary Rehabilitation Program vs Tai Chi + PRP; power of 0.80 for medium effect size at 5% level of significance; Test type: Superiority or Other; p = 0.528, ANCOVA; adjusted for baseline value, age, sex, BMI, education and smoking; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-3.5 to 6.8], Standard Deviation 5.2

ADVERSE EVENTS:
Time Frame: Both PRP and PRP+Tai chi were followed up to 6 months post-intervention.
Description: "serious" and "other " adverse events were not assessed and collected
Groups:
- PRP + Tai Chi: Tai Chi elements added to PRP program
- Pulmonary Rehabilitation Program PRP: Subjects who received formal pulmonary rehabilitation program
Arm/Group | PRP + Tai Chi | Pulmonary Rehabilitation Program PRP
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
There was high attrition rate of 28% which further contributed to our small sample size with wide 95% confidence interval of several outcome variables results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No